CLINICAL TRIAL: NCT04168723
Title: A Phase 1, Single-Center, Double-Blind, Randomized, Placebo- and Positive Controlled, Double-Dummy, Parallel-Group, Repeated Dose Study With a Nested Cross-Over Comparison Between Moxifloxacin and Placebo to Evaluate the Effect of MD1003 on Cardiac Repolarization in Healthy Adult Subjects
Brief Title: TQT2 Study to Evaluate the Effect of MD1003 on Cardiac Repolarization in Healthy Adult Subjects
Acronym: TQT2
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MedDay Pharmaceuticals SA (Industry)
Collaborators: Parexel (Industry); ERT: Clinical Trial Technology Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MD1003CT2019-04TQT2
Record Dates: First submitted 2019-11-08; First posted 2019-11-19 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Biotin; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Double-Blind, Randomized, Placebo- and Positive Controlled, Double-Dummy, Parallel-Group, Repeated-Dose Study with a Nested Cross-Over Comparison Between Moxifloxacin and Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A-MD1003 (Experimental): Group A=32 subjects Placebo for MD1003 on Day -1. Daily dose of 1200 mg of MD1003 from Day 1 to Day 8 Placebo for moxifloxacin on Day 1 and Day 9
  Interventions: Drug: MD1003; Drug: Placebo for MD1003; Drug: Placebo for moxifloxacin
- Group B-Moxifloxacin (Active Comparator): Subjects in Group B will be further randomized to Subgroups B1 and B2 in a ratio of 1:1.
  Subgroup B1: 16 subjects Placebo for MD1003 on Day -1 Placebo for MD1003 from Day 1 to Day 8 Moxifloxacin 400 mg on Day 1 and Placebo for moxifloxacin on Day 9 Subgroup B2: 16 subjects Placebo for MD1003 on Day -1 Placebo for MD1003 from Day 1 to Day 8 Placebo for moxifloxacin on Day 1 and Moxifloxacin 400 mg on Day 9
  Interventions: Drug: Moxifloxacin 400mg; Drug: Placebo for MD1003; Drug: Placebo for moxifloxacin

INTERVENTIONS:
Drug: MD1003 — Group A: Daily dose of 1200 mg of MD1003 from Day 1 to Day 8
  Other Names: Biotin
  Arms: Group A-MD1003
Drug: Moxifloxacin 400mg — Group B1: Moxifloxacin 400 mg on Day 1 Group B2: Moxifloxacin 400 mg on Day 9
  Other Names: Moxifloxacin
  Arms: Group B-Moxifloxacin
Drug: Placebo for MD1003 — Group A: Placebo for MD1003 on Day -1 Group B1: Placebo for MD1003 on Day -1 Group B2: Placebo for MD1003 on Day -1
Drug: Placebo for moxifloxacin — Group A: Placebo for moxifloxacin on Day 1 and Day 9 Group B1: Placebo for moxifloxacin on Day 9 Group B2: Placebo for moxifloxacin on Day 1

SUMMARY:
This is a Phase 1, single-center, double-blind, randomized, placebo- and positive controlled, double-dummy, parallel-group, repeated-dose study with a nested cross-over comparison between moxifloxacin and placebo to evaluate the effect of MD1003 on cardiac repolarization in healthy adult subjects.

The planned enrollment is approximately 64 subjects randomized in a ratio of 1:1 to 2main groups. Subjects in Group B will be further randomized to Subgroups B1 and B2 in a ratio of 1:1.

DETAILED DESCRIPTION:
This study is designed as a definitive evaluation of the potential of MD1003 and its major metabolites to have a threshold effect on cardiac repolarization, as detected by QT/QTc prolongation. The design is aligned with the recommendations for evaluation of QT/QTc interval prolongation outlined in the International Council for Harmonization (ICH) E14 guidance.

This is a Phase 1, single-center, double-blind, randomized, placebo- and positive controlled, double-dummy, parallel-group, repeated-dose study with a nested cross-over comparison between moxifloxacin and placebo to evaluate the effect of MD1003 on cardiac repolarization in healthy adult subjects.

A total of 64 subjects will be enrolled in the clinical study according to the inclusion/exclusion criteria. The study consists of two main groups with 32 subjects per dose group. All subjects will receive placebo for MD1003 on Day -1. Subjects in Group A will receive MD1003 (biotin) 1200 mg and placebo for moxifloxacin on Day 1, MD1003 (biotin) 1200 mg from Day 2 through Day 8 and placebo for moxifloxacin on Day 9. Subjects in Group B will be further randomized to Subgroup B1 (16 subjects) receiving moxifloxacin 400 mg and placebo for MD1003 on Day 1, placebo for MD1003 from Day 2 through Day 8 and placebo for moxifloxacin on Day 9. Subgroup B2 (16 subjects) will receive placebo for moxifloxacin and placebo for MD1003 on Day 1, placebo for MD1003 from Day 2 through Day 8 and moxifloxacin 400 mg on Day 9.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent form prior to performing any of the Screening Visit procedures.
2. Males and females between 18 to 55 years of age, inclusive, at the Screening Visit.
3. Female subjects of childbearing potential must not be planning to become pregnant, must not be breastfeeding, and must have a negative serum pregnancy test at Screening and negative urine pregnancy test on Day-2.
4. Sexually active female subjects of childbearing potential (i.e. women who are not post-menopausal [12 months of spontaneous amenorrhea without an alternative medical cause and follicle stimulating hormone (FSH) levels in the post-menopausal range for the laboratory involved] or who have not had a documented hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) and all male subjects (who have not been surgically sterilized by documented vasectomy) must agree to use highly effective methods of contraception during the study and for 8 weeks after the last dose of study drug. Please refer to Section 5.4.4 for acceptable methods of contraception.
5. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the screening.
6. Body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive, at the Screening Visit.
7. Healthy adult subjects with suitable veins for cannulation.
8. Healthy, determined by pre-study medical evaluation (medical history, renal function, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations).
9. Supine vital signs should be within the normal range at Screening and Day -2:

   1. oral body temperature between 35.0°C - 37.5°C;
   2. systolic BP, 90 - 140 mm Hg;
   3. diastolic BP, 40 - 90 mm Hg;
   4. pulse rate, 40 - 100 bpm.
10. Subjects should have serum potassium, calcium, and magnesium levels within the normal range at Screening and at admission on Day -2 (morning in fasted condition).
11. Subjects should fulfil the following ECG parameters criteria at Screening and Day -2:

    1. Normal sinus rhythm (HR between 40 beats per minute [bpm] and 100 bpm, inclusive);
    2. Fridericia QTc interval corrected (QTcF)≤ 450 msec;
    3. QRS interval ≤110 msec; and confirmed by manual over-read if > 110 msec;
    4. PR interval ≤220 msec.

Exclusion criteria:

1. Subject has clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological or psychiatric disorder(s) as determined by the Principal Investigator or designee.
2. Subject has any disorder that would interfere with the absorption, distribution, metabolism or excretion of drugs.
3. Subject has any concurrent disease or condition that, in the opinion of the Principal Investigator, would make the subject unsuitable for participation in the clinical study.
4. History or presence of:

   1. risk factors for Torsades de Pointes (e.g., heart failure, cardiomyopathy, or family history of Long QT Syndrome);
   2. sick sinus syndrome, Mobitz 2second, or third-degree atrioventricular block, myocardial infarction, pulmonary congestion, cardiac arrhythmia, prolonged QT interval QTc>450 male/470 female), or conduction abnormalities;
   3. repeated or frequent syncope or vasovagal episodes;
   4. hypertension, angina, bradycardia, or severe peripheral arterial circulatory disorders.
5. Subjects with serum creatinine clearance below 90 mL/min.
6. Subject has history of alcohol and/or illicit drug abuse within 2 years prior to the first dose of study drug.
7. Subject has positive test for Hepatitis B surface antigen, Hepatitis C antibody or human immunodeficiency virus antibody at the screening visit.
8. Subject has positive urine drug (e.g., cocaine, amphetamines, barbiturates, opiates, benzodiazepines, cannabinoids), alcohol or cotinine test at the Screening Visit or Day -2. Consumption of alcohol and alcohol-containing foods, medications or beverages 48 hours prior to the screening visit.
9. Female subjects are breastfeeding or female subjects with a positive serum pregnancy test at the Screening Visit or positive urine pregnancy test on Day -2.
10. Has had surgery or any medical condition which may affect the absorption, distribution, metabolism, or elimination of the study drugs within 6 months prior to the first dose, in the opinion of the Principal Investigator.
11. Plasma donation within 7 days prior to the first dose of study drug.
12. Subject has donated > 500 mL blood or blood products within 2 months (56 days) prior to admission.
13. Subject is unwilling to avoid consumption of coffee and caffeine containing beverages from 48 hours prior to admission until discharge from the clinical site.
14. Use of any prescription or over-the-counter medication including antacids, herbal remedies, or vitamin or nutritional supplements (especially those containing biotin, magnesium, aluminum, iron, or zinc), excluding contraceptive pill, and intermittent use of paracetamol, ibuprofen, or acetylic salicylic acid within 14 days prior to Screening and throughout the study, unless approved by both the Investigator and the Sponsor.
15. Subject has used an investigational drug, or device within 3 months or 5 half-lives of the investigational drug (whichever is longer) prior to Screening.
16. Participation in a previous clinical trial where subject received MD1003.
17. Subject has been on a diet incompatible with the on study diet (including an extreme diet which resulted in a significant weight change for whatever reason), in the opinion of the Principal Investigator, within the 28 days prior to the first dose of study drug, and throughout the study.
18. Subject is unwilling to abstain from vigorous exercise from 48 hours prior to admission until the End of Study Visit.
19. Subject has a history of hypersensitivity to the study drug or any of the excipients (incl. lactose), or to medicinal products with similar chemical structures.
20. Subject is unlikely to comply with the protocol requirements, instructions and study related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits and improbability of completing the clinical study.
21. Vulnerable subjects defined as individuals whose willingness to volunteer in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate (e.g., persons in detention, minors and those incapable of giving consent).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-03-05 (Estimated); Study Completion 2020-03-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline QTcF (ΔQTcF) on Day 8 (after 8 days of 1200 mg MD1003) | 9 days
  Replicate electrocardiograms (ECGs) (10 ECG replicates) for the determination of ΔQTc interval will be extracted from the continuous digital 12-lead ECG recording in the 5 minutes prior to dosing and then at 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose on D-1 and D8

SECONDARY OUTCOMES:
Placebo-corrected change from baseline QTcF (ΔΔQTcF) on Day 8 (after 8 days of 1200 mg MD1003) | 9 days
  Replicate electrocardiograms (ECGs) (10 ECG replicates) for the determination of ΔΔQTc interval will be extracted from the continuous digital 12-lead ECG recording in the 5 minutes prior to dosing and then at 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose on D-1 and D8
Change from baseline of Heart Rate (ΔHR) on Day 8 (after 8 days of 1200 mg MD1003) | 9 days
  Replicate electrocardiograms (ECGs) (10 ECG replicates) for the determination of ΔHR interval will be extracted from the continuous digital 12-lead ECG recording in the 5 minutes prior to dosing and then at 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose on D-1 and D8
Placebo-corrected, change from baseline of Heart Rate (ΔΔHR) on Day 8 (after 8 days of 1200 mg MD1003) | 9 days
  Replicate electrocardiograms (ECGs) (10 ECG replicates) for the determination of ΔΔHR interval will be extracted from the continuous digital 12-lead ECG recording in the 5 minutes prior to dosing and then at 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose on D-1 and D8
Change from baseline of Pulse Rate (ΔPR) on Day 8 (after 8 days of 1200 mg MD1003) | 8 days
  Measurement of PR will be performed manually in 3 of the 9 ECG replicates at each timepoint at 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose on D1 and D8
Placebo-corrected, change from baseline of Pulse Rate (ΔΔPR) on Day 8 (after 8 days of 1200 mg MD1003) | 8 days
  Measurement of PR will be performed manually in 3 of the 9 ECG replicates at each timepoint at 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose on D1 and D8
Change from baseline of QRS interval (ΔQRS) on Day 8 (after 8 days of 1200 mg MD1003) | 8 days
  Measurement of QRS interval will be performed manually in 3 of the 9 ECG replicates at each timepoint at 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose on D1 and D8
Placebo-corrected, change from baseline of QRS interval (ΔΔQRS) on Day 8 (after 8 days of 1200 mg MD1003) | 8 days
  Measurement of QRS interval will be performed manually in 3 of the 9 ECG replicates at each timepoint at 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose on D1 and D8
T-wave morphology | 8 days
  Frequency of treatment emergent changes in T-wave morphology. Measurement of T-wave morphology will be performed manually in 3 of the 9 ECG replicates at each timepoint at 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose on D1 and D8
U-waves presence | 8 days
  Frequency of treatment emergent changes in U-waves presence. Measurement of U-waves presence will be performed manually in 3 of the 9 ECG replicates at each timepoint at 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose on D1 and D8
Maximum plasma concentrations (Cmax) of MD1003 will be measured at D1 and D8 post-dose (after 8 days of dosing of 1200mg of MD1003) | 8 days
  The measured individual plasma concentration at pre-dose then at 0.5, 1, 2, 3, 4, 8,12, 24 hours (D1 and D8) post-dose will be used to directly obtain Cmax. Unit: ng/ml.
Area under the curve (AUC max) of MD1003 will be measured at D1 and D8 post-dose (after 8 days of dosing of 1200mg of MD1003) | 8 days
  AUC max at pre-dose then at 0.5, 1, 2, 3, 4, 8,12, 24 hours (D1 and D8) post-dose will be used to directly obtain AUC max. Unit: ng.h/ml
Time for maximum plasma concentration (tmax) of MD1003 will be determined directly from the concentration-time profile | 8 days
  tmax will be determined directly from the concentration-time profile. Unit: hour

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, MD, Principal Investigator — Parexel Early Phase Clinical Unit London,Northwick Park Hospital
Locations (1):
- Parexel Early Phase Clinical Unit London, London, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No